CLINICAL TRIAL: NCT00690404
Title: A Phase 1, Single-center, Randomized, Open-label, Two-way Crossover, Formulation and Food Effect Study in Healthy Volunteers, to Assess the Pharmacokinetics of AZD 2066 After Single Doses of a New Oral Solid Formulation and an Oral Solution
Brief Title: AZD 2066 Single Dose Formulation and Food Effect Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Rolf Karlsten, M.D., Medical Science Director, Emerging Neuroscience, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: D0475C00005
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: formulation; pharmacokinetic; crossover formulation; food effect; oral solution; healthy volunteers
MeSH Terms: interventions — AZD2066

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD2066

INTERVENTIONS:
Drug: AZD2066 — single oral dose

SUMMARY:
A open label two way crossover formulation and food effect study in healthy volunteers to assess the pharmacokinetics of a single dose of AZD2066 new oral solid formulation and an oral solution

ELIGIBILITY:
Inclusion Criteria:

* Clinical normal physical findings, including BP, pulse rate >45 bpm, ECG and laboratory assessments
* Body Mass Index (BMI) of ≥18 to ≤30 kg/m2 and weight of ≥50 to ≤100 kg

Exclusion Criteria:

* History of hypersensitivity, allergy or atopic/skin disease as judged by Investigator.
* History of somatic or psychiatric disease/condition, which may interfere with the objectives of the study as judged by the Investigator.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
AZ2066 pharmacokinetics | several samples within 72 hrs

SECONDARY OUTCOMES:
Effect of food on AZD2066 pharmacokinetics | several samples over 72 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Lisbon, MD, MPH, Principal Investigator — Quintiles, Inc. Overland Park, Kansas, USA; Heather Wray, MB, ChB, FFPM, Study Chair — AstraZeneca Charnwood England; Ivan Eggens, MD, Study Chair — AstraZeneca , Södertälje, Sweden